CLINICAL TRIAL: NCT03529279
Title: CNG Staging Compared With UICC Eighth Staging of Nasopharyngeal Carcinoma for Treatment Decision-marking and Selection of Chemotherapy and Radiotherapy： a Multicenter, Open Label, Randomized Controlled, Non-inferiority Clinical Trial
Brief Title: CNG Staging Compared With 8th UICC of NPC for Treatment Decision-marking and Selection of Chemotherapy and Radiotherapy
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yun-fei Xia, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B2018-030-01
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The patients in the Experimental Group are allocated to receive CNG staging and CNG chemotherapy strategy and CNG radiation strategy
  Interventions: Drug: CNG Chemotherapy; Radiation: CNG Radiation
- Controlled Group (Active Comparator): The patients in the Controlled Group are allocated to receive the eighth edition of UICC/AJCC staging and NCCN chemotherapy strategy and NCCN radiation strategy
  Interventions: Drug: NCCN Chemotherapy; Radiation: NCCN Radiation

INTERVENTIONS:
Drug: CNG Chemotherapy — CNG I, IMRT plus oral adjuvant chemotherapy, if EBV-DNA > 0,according to CNG II. CNG II, IMRT + concurrent chemotherapy + oral adjuvant chemotherapy. CNG III, systemic chemotherapy, plus IMRT.
  Chemotherapy strategy: Concurrent chemotherapy, 5-Fu + nedaplatin (cisplatin), every 28 days; 5-Fu 500mg/m2. D, civ d1-d5, nedaplatin (cisplatin) 80mg (70mg) /m2. D, D1. Systemic chemotherapy, 5-Fu + nedaplatin (cisplatin), every 60 days; 5-Fu (100 - 200 mg/m2. D) civ for 30 days, nedaplatin (cisplatin) 80mg (70mg) /m2. D, D1,D28. Aim to achieve CR in imaging.Oral adjuvant chemotherapy, tegafon (400 mg, QID) and Calcium Folinate Tablets (30 mg, QID). Oral 10 days and stop 20 days, 3 months/course. After 6 courses, oral 10 days and stop 50 days, half year/course, 6-7 courses, lasted for 5 years.
  Other Names: Chemotherapy strategy for experimental group
  Arms: Experimental Group
Drug: NCCN Chemotherapy — UICC I, IMRT. UICC II-IVA, concurrent chemoradiotherapy ± adjuvant chemotherapy, or induced chemotherapy plus concurrent chemoradiotherapy. UICC IVB, platinum based combined chemotherapy, followed by IMRT or concurrent chemoradiotherapy, or concurrent chemoradiotherapy.
  Chemotherapy strategy: Concurrent cisplatin with or without cisplatin plus 5-Fu or carboplatin combined with 5-Fu adjuvant chemotherapy; The combined chemotherapy regimen of IVB stage patients may choose cisplatin or carboplatin plus docetaxel or paclitaxel, cisplatin plus 5-Fu, carboplatin and cetuximab, cisplatin plus gemcitabine, and gemcitabine. The combination of vinorelbine and cisplatin, carboplatin, paclitaxel, docetaxel, 5-Fu, methotrexate, gemcitabine and capecitabine can be used in combination with radiotherapy.
  Other Names: Chemotherapy strategy for controlled group
  Arms: Controlled Group
Radiation: CNG Radiation — IMRT technique. GTV was given to 6810cGy, CTV1 was given to 6000cGy, and CTV2 was given to 4800-5400cGy. 30 fractions, daily, QW1-5.
  CT-SIM or MR-CIM was evaluated every 10 fractions. If CR for CNG I and II patients at 10 fractions, radiotherapy were given 25 fractions, that was, GTV was given to 5675cGy, CTV1 was given 5000cGy, and CTV2 was given 4000-4500cGy, 25 fractions, daily, QW1-5.
  If tumor reduced less than 50% at 20 fractions, GTV was modified according to tumor size at 20 fractions. The modified GTV was given 300cGy/F×5 after 25 fractions; the original CTV1 and CTV2 were unchanged, that is, GTV was given to 5675cGy/25Fr+1500cGy/5Fr and CTV1 was given to 6000cGy/30Fr, CTV2 was given 4800-5400cGy/30Fr.
  Other Names: Radiation for experimental group
  Arms: Experimental Group
Radiation: NCCN Radiation — IMRT technique. When IMRT alone, GTV were given (1) 66Gy (2.2Gy/Fr) to 70-70.2 Gy (1.8-2.0 Gy/Fr), QW1-5, 6-7 weeks; (2) 69.96 Gy (2.12 Gy/Fr), 6-7 weeks; CTV1-2 were given 44-50 (2.0 Gy/Fr) to 54-63 (1.8 Gy/Fr).
  When combined with chemotherapy, GTV were given 70-70.2 Gy (1.8-2.0 Gy/Fr), QW1-5, 7 weeks; CTV1-2 were given 44-50 Gy (2 Gy/Fr) to 54-63 Gy (1.8 Gy/Fr).
  When palliative radiotherapy, 50Gy/20Fr; 37.5 Gy/15Fr (if tolerable, increases 5 fractions to 50Gy); 30Gy/10Fr, 30Gy/5Fr, 2 fractions per week, interval more than 3 days; 44.4Gy/12Fr was divided into 3 cycles, 2 fractions a day, 6 hours of interval, 2 consecutive days and 3-4 weeks between two cycles. After second cycles, the treatment plan must completely avoid the irradiation of the spinal cord.
  Other Names: Radiation for controlled group
  Arms: Controlled Group

SUMMARY:
Due to the increase of tumor control rate and survival rate in era of IMRT, the role of the seventh edition of UICC/AJCC staging system in predicting prognosis is becoming weaker and inaccurate.

Therefore, we put forward a new staging for the clinical staging of NPC in the era of IMRT without changing the current T, N, M staging definition of the 7th of the UICC/AJCC staging system. We call this new stage "Cooperative Nasopharyngeal Carcinoma Group" stage, namely CNG stage. In CNG stage, the clinical stages were reduced to three stages, namely, CNG I stage includes T1-3N0-1M0 and T1-2N2M0, CNG II stage includes T3N2M0, T4N0-2M0 and TanyN3M0, CNG III stage includes TanyNanyM1. For CNG I stage, the IMRT alone is sufficient. If EBV-DNA copies is more than 0 copy/ml, concurrent chemoradiotherapy will be given. For CNG II stage, patients can benefit from combined radiotherapy and chemotherapy. For CNG III stage, patients are recommended for systemic chemotherapy plus local radiotherapy (primary focus, neck drainage area and distant metastasis).

This year, UICC/AJCC has proposed an eighth edition of NPC staging system. The eighth version is mainly changed in the definition and refinement of the anatomic location compared with the seventh edition. This is different from our new CNG staging concept.

Therefore, CNG staging and its treatment strategy was used as the experimental group, and the eighth edition of UICC/AJCC staging with NCCN guiding treatment was used as the control group. The open and randomized controlled clinical study was conducted. The purpose of this study was to evaluate in the era of IMRT, CNG staging can be better than UICC/AJCC eighth clinical staging for treatment decision-marking and selection of chemotherapy and radiotherapy, and differentiating differences in prognosis in each clinical stage. The survival results based on CNG staging and its treatment are not inferior to the survival results of the NCCN guide therapy based on the eighth edition UICC/AJCC staging, to avoid chemotherapy for some of the patients, and to improve the outcome of metastatic patients.

DETAILED DESCRIPTION:
The seventh edition of the UICC/AJCC staging system, which is widely used in recent years, is based on survival data in the traditional era of radiotherapy. However, the survival of nasopharyngeal cancer patients has been greatly improved in the era of modern radiation therapy, which IMRT (Intension Modulated Radiotherapy) is widely used. Even with radiotherapy alone, the 5 year disease specific survival rate of nasopharyngeal carcinoma with stage I-II is more than 95%, the 3 year overall survival rate of non metastatic III-IV patients is about 75%, and the 5 year overall survival rate is about 80%. The 5 year survival rate of metastatic nasopharyngeal carcinoma can reach more than 20% with systemic treatment. Due to the increase of tumor control rate and survival rate in era of IMRT, the role of the seventh edition of UICC/AJCC staging system in predicting prognosis is becoming weaker and inaccurate.

Therefore, in the previous study, we put forward a new staging for the clinical staging of nasopharyngeal carcinoma in the era of IMRT without changing the current T, N, M staging definition of the seventh edition of the UICC/AJCC staging system. We call this new stage "Cooperative Nasopharyngeal Carcinoma Group" stage, namely CNG stage. In CNG stage, the clinical stages were reduced to three stages, namely, CNG I stage includes T1-3N0-1M0 and T1-2N2M0, CNG II stage includes T3N2M0, T4N0-2M0 and TanyN3M0, CNG III stage includes TanyNanyM1, and the 5 year DSS (Disease specific survival) is 93.3%, 72.7%, and 24%, respectively, with a significant difference.

This year, UICC/AJCC has proposed an eighth edition of nasopharyngeal carcinoma staging system based on the revision of the seventh edition. The main updates are: (1) add the definition of the T0 phase, that is, the EBV positive cervical lymph node metastases with uncertain primary foci, and (2) the invasion of the adjacent muscles (including the pterygus, the extradypterygus, and the anterior vertebroid muscle) into T2; (3) replace the "masticatory muscle space" and "subtemporal fossa" in the previous T4 definition with a specific description of soft tissue invasion; (4) change the supraclavicular fossa to the lower neck (defined as the lymph node metastases below the subchondral edge); (5) N3a and N3b are combined called N3, and it is defined as a single / double neck lymph node with long diameter > 6cm, and/or below the subchondral subchondral edge; (6) the IVA stage (T4 N0-2 M0) and the IVB stage (anyT N3 M0) are combined called IVA stage; (7) the IVC stage (anyT anyN) is changed to IVB stage. The eighth version is mainly changed in the definition and refinement of the anatomic location compared with the seventh edition. Except for the migration of the adjacent muscle invasion, and the other changes are not significant. The upper bound of N3 is moved from the supraclavicular fossa to the subchondral edge in N staging. This is different from our new CNG staging concept.

CNG staging of nasopharyngeal carcinoma is related to the unique biological behavior of nasopharyngeal carcinoma, which is consistent with the three clinical patterns of nasopharyngeal carcinoma, namely, non metastasis, tendency to metastasis and metastasis. The pattern of tendency to metastasis was related to the late T and N staging. Based on the biological behavior and clinical survival data of NPC, we further proposed the treatment strategy of nasopharyngeal carcinoma under the guidance of CNG staging, that is, the CNG I stage is consistent with the non metastasis model, and the IMRT alone is sufficient. The CNG II stage is consistent with the tendency to metastasis mode, which can benefit from combined radiotherapy and chemotherapy. The CNG III stage is metastatic mode, which is recommended for systemic chemotherapy plus local radiotherapy (primary focus, neck drainage area and distant metastasis). In clinical practice, we suggest that for patients with CNG I stage, if EBV-DNA copies is more than 0 copy/ml, concurrent chemoradiotherapy will be given.

Therefore, CNG staging and its treatment strategy was used as the experimental group, and the eighth edition of UICC/AJCC staging with NCCN guiding treatment was used as the control group. The open and randomized controlled clinical study was conducted. The purpose of this study was to evaluate in the era of IMRT, CNG staging can be better than UICC/AJCC eighth clinical staging for treatment decision-marking and selection of chemotherapy and radiotherapy, and differentiating differences in prognosis in each clinical stage. The survival results based on CNG staging and its treatment are not inferior to the survival results of the NCCN guide therapy based on the eighth edition UICC/AJCC staging, to avoid chemotherapy for some of the patients, and to improve the outcome of metastatic patients.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed and previously untreated nasopharyngeal carcinoma
* Non T1N0M0 patient according to UICC/AJCC seventh edition staging system
* Age ≥ 18 years and < 65 years
* Karnofsky performance status (KPS) score ≥ 70
* Adequate normal organ function
* No history of other malignant tumors
* No serious mental disorder (schizophrenia, delusion of victimization, manic depression, and drug induced anxiety)
* No AIDS, active pulmonary tuberculosis and other serious immunodeficiency diseases
* No communication barrier, can answer the question
* Sign informed consent under voluntary circumstances, complete treatment and follow up as required

Exclusion Criteria:

* Poor compliance
* Investigators consider as inappropriate for enrolling into this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1324 (Estimated)
Dates: Start 2018-06-12 (Estimated); Primary Completion 2026-06-12 (Estimated); Study Completion 2026-06-12 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From the date of randomization until the date of death, assessed up to 60 months
  5-year overall survival

SECONDARY OUTCOMES:
Quality of life | From the date of radiotherapy begin, every week during radiotherapy, assessed up to 60 months
  The standard scores assessed by EORTC QOL scale decreased by more than 10 points
Recurrence free survival (RFS) | From the date of randomization until the date of first recurrence, assessed up to 60 months
  5-year recurrence free survival
Distant metastasis free survival (DMFS) | From the date of randomization until the date of first distant metastasis, assessed up to 60 months
  5-year distant metastasis free survival
Disease specific survival (DSS) | From the date of randomization until the date of death from tumor, assessed up to 60 months
  5-year disease specific survival
Complete remission (CR) | From the date of randomization, 3 months after radiotherapy
  all the target lesions disappeared, no new lesions appeared, and the tumor markers were normal, and maintained for at least 4 weeks, according to RECIST
Incidence of side effects associated with tumor therapy | From the date of randomization up to 60 months
  according to NCI CTC 4.0

CONTACTS AND LOCATIONS:
Overall Officials: Yun-fei Xia, M.D, Principal Investigator — Sun Yat-sen University

REFERENCES:
- [Derived] Zheng S, Liu Y, He Z, He S, Huang Z, Luo W, Han F, Tao Y, Chen C, Ouyang P, Chen L, Huang Y, Zhou G, Li W, Liu Q, Chen C, Xia Y. CNG (Collaborative Nasopharyngeal Carcinoma Group) stage: Improved prognostic stratification of nasopharyngeal carcinoma and association with Epstein-Barr virus DNA in the intensity-modulated radiation therapy era. Radiother Oncol. 2025 Sep;210:111051. doi: 10.1016/j.radonc.2025.111051. Epub 2025 Jul 19. PMID 40692079